CLINICAL TRIAL: NCT00046761
Title: A Study to Evaluate the Effects of ONO-2506 Intravenous Infusion in Patients With Acute Ischemic Stroke
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2506/INT0104
Record Dates: First submitted 2002-10-02; First posted 2002-10-04 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Cerebrovascular Accident
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — ONO2506

INTERVENTIONS:
Drug: ONO-2506

SUMMARY:
The primary objective of this study is to compare the efficacy of ONO-2506 versus placebo in neurological stroke outcome in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a clinical diagnosis of acute cortical ischemic stroke.
* Patient must be randomized into the study within six hours after the initial onset of stroke symptoms.
* Patient must have a measurable focal neurological deficit for a minimum duration of 60 minutes.
* Patient must have a CT or MRI examination compatible with the clinical diagnosis of acute ischemic stroke.
* Patient must have had a pre-stroke mRS scale score of 0 or 1.
* Other inclusion criteria as specified in the study protocol.

Exclusion Criteria:

* Patient must not have a body weight of more than 125 kg.
* Patient must not have a CT and/or MRI with evidence of a non-ischemic mechanism, subarachnoid hemorrhage, or primary intracerebral and/or intraventricular hemorrhage.
* Patient must not have all three of the following findings:

  1. reduced level of consciousness (has score of greater than or equal to two on NIHSS Question 1a)
  2. forced eye deviation or total gaze paresis (has score of 2 on NIHSS Question 2) and
  3. dense hemiplegia (no movement) of upper and lower extremities (i.e., has score of 4 on NIHSS Question 5 regarding motor arm and has score of 4 on NIHSS Question 6 regarding motor leg).
* Patient must not have neurological signs and symptoms that are rapidly improving.
* Patient must not have a severe coexisting or terminal systemic disease.
* Patient must not be pregnant or lactating.
* Patient must not have impaired hepatic function; bilirubin greater than 2 mg/dL and or ascites.
* Patient must not have impaired renal function; serum creatinine greater than 2 mg/dL.
* Patient must not have congestive heart failure.
* Patient must not have a baseline ECG showing a PR interval greater than 200 milliseconds, or a corrected QT interval of greater than 480 milliseconds, or a history of ventricular arrhythmias, or a Mobitz Type 1 or greater AV block.
* Patient must not have other exclusion criteria as specified in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320
Dates: Start 2002-11; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Due, Ph.D., Study Director — Ono Pharma USA Inc
Locations (148):
- United States (130):
  - Brookwood Medical Center, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - Alta Bates Hospital/ Summit Medical Center, Berkeley, California
  - Grossmont Hospital, La Mesa, California
  - Loma Linda University Medical Center, Loma Linda, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford Stroke Center, Palo Alto, California
  - Mercy Medical Center, Redding, California
  - Redding Medical Center, Redding, California
  - UC Davis Medical Center, Sacramento, California
  - Good Samaritan Hospital, San Jose, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - The Stroke Center at Hartford Hospital, Hartford, Connecticut
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - North Broward Medical Center, Fort Lauderdale, Florida
  - Alachua General Hospital, Gainsville, Florida
  - Aventura Hospital and Medical Center, Hollywood, Florida
  - Neurology Associates, PA, Maitland, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Ocala Regional Medical Center, Ocala, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - BonSecours - St. Joseph's Hospital, Port Charlotte, Florida
  - Charlotte Regional Medical Center, Port Charlotte, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Palms of Pasadina Hospital, St. Petersburg, Florida
  - St. Joseph Hospital, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - Memorial Hospital of Tampa, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - St. Francis Hospital, Columbus, Georgia
  - DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Decatur, Georgia
  - Joan Glancy Memorial Hospital, Decatur, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - MacNeal Hospital, Berwyn, Illinois
  - BroMenn Regional Medical Center, Bloomington, Illinois
  - OSF St. Joseph Medical Center, Bloomington, Illinois
  - Alexian Brothers Hospital, Elk Grove Village, Illinois
  - Advocate Christ Hospital & Medical Center, Oak Lawn, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Central DuPage Hospital, Warrenville, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - Parkview Hospital, Fort Wayne, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lexington Clinic, Lexington, Kentucky
  - Chandler Medical Center /Univ of Kentucky, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Detroit Receiving Hospital/ Wayne State Univ, Detroit, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. John's Clinic - Smith-Glynn-Callaway, Springfield, Missouri
  - Benefits Healthcare/ Advanced Neurology Specialists, Great Falls, Montana
  - Creighton University Medical Center, Omaha, Nebraska
  - Washoe Medical Center, Reno, Nevada
  - Cooper Hospital /University Medical Center, Camden, New Jersey
  - JFK Medical Center, Edison, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Virtua Memorial Hospital, Medford, New Jersey
  - Robert Wood Johnson Hospital, New Brunswick, New Jersey
  - Muhlenberg Hospital, Plainfield, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - St. Peter's Hospital, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - Millard Fillmore Hospital, Buffalo, New York
  - Wilson Memorial Regional Medical Center, Johnson City, New York
  - North Shore University Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Vernon Hospital, Mount Vernon, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mt. Sinai Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York
  - Ellis Hospital Stroke Center B421, Schenectady, New York
  - SUNY Stony Brook University Hospital, Stony Brook, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Kettering Medical Center -Wallace Kettering Neuroscience Inst., Kettering, Ohio
  - Medical College of Ohio Hospital, Toledo, Ohio
  - St. Elizabeth's Health Center, Youngstown, Ohio
  - Rogue Valley Medical Center, Medford, Oregon
  - Oregon Health and Science University - Oregon Stroke Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent's Hospital, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Crozer Chester Medical Center, Upland, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Greenville Hospital, Greenville, South Carolina
  - Erlanger Hospital, Chattanooga, Tennessee
  - Regional Medical Center at Memphis, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas; Southwestern Medical Center at Dallas, Dallas, Texas
  - Methodist Hospital /Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University Hospital /Univ of Texas Health Science Center, San Antonio, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - The Innovative Clincal Research Center, Alexandria, Virginia
  - Virginia Commonwealth University /Medical College of VA, Richmond, Virginia
  - Henrico Doctors Hospital, Richmond, Virginia
  - Memorial Regional Medical Center, Richmond, Virginia
  - St. Mary's Hospital, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - St. Joseph's Hospital/ Marshfield Clinic, Marshfield, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Theda Clark Medical Center, Neenah, Wisconsin
- Canada (18):
  - Foothills Medical Center /University of Calgary, Calgary, Alberta
  - University of Alberta Hospital /Mackenzie Center, Edmonton, Alberta
  - Lethbridge Regional Hospital, Lethbridge, Alberta
  - Royal Inland Hospital, Kamloops, British Columbia
  - Kelowna General Hospital, Kelowna, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - York Central Hospital, Richmond Hill, Ontario
  - Complexe Hospitalier de La Sagamie, Chicoutimi, Quebec
  - Centre Hospitalier des Vallees de l'Outaouais, Gatineau, Quebec
  - Hotel-Dieu de Levis, Lévis, Quebec
  - Hospital Notre Dame du Chum, Montreal, Quebec
  - Hotel-Dieu de St-Jerome, Saint-Jérôme, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan